CLINICAL TRIAL: NCT07033481
Title: A Phase 2a Clinical Study of the P38 Alpha Kinase Inhibitor Neflamapimod in Patients With Primary Progressive Aphasia (PPA)
Brief Title: Clinical Study of Neflamapimod in Patients With Primary Progressive Aphasia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: EIP Pharma Inc (Industry)
Collaborators: CervoMed, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRVO24-NFD-701
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Nonfluent Variant Primary Progressive Aphasia (nfvPPA)
Keywords: Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Neurocognitive Disorders; Mental Disorders; Neurodegenerative Diseases; Aphasia; Language Disorder; Frontotemporal Dementia; Speech and Language Disorder; Primary Progressive Aphasia
MeSH Terms: conditions — Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Neurocognitive Disorders; Mental Disorders; Neurodegenerative Diseases; Aphasia; Language Disorders; Frontotemporal Dementia; Speech; Aphasia, Primary Progressive

STUDY DESIGN:
Intervention Model Description: All participants will be assigned 40 milligram (mg) neflamapimod three times per day (TID) for 24 weeks. Following completion of the 24-week open-label treatment period, participants will continue to a randomized, double-blinded withdrawal period and be randomly assigned on a 1:1 basis to neflamapimod or placebo for 12 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neflamapimod (Experimental)
  Interventions: Drug: Neflamapimod
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Neflamapimod — Neflamapimod is a highly specific inhibitor of the intra-cellular enzyme mitogen-activated protein kinase14 (p38α) provided in 40 mg capsules
  Arms: Neflamapimod
Drug: Placebo — Placebo is a capsule that looks just like neflamapimod but without the active ingredients
  Arms: Placebo

SUMMARY:
The goal of this exploratory study is to evaluate the effect of neflamapimod in participants with nonfluent variant primary progressive aphasia (nfvPPA). We aim to evaluate the safety, pharmacokinetics and clinical effects of neflamapimod of participants with nfvPPA.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 40-85 years at Screening.
* Participant or participant's legally authorized representative (where applicable) is willing and able to provide written informed consent.
* Clinical diagnosis of nfvPPA by consensus criteria [Gorno-Tempini et al, 2011].

  * At least one of the following core features must be present:

    1. Agrammatism in language production
    2. Effortful, halting speech with inconsistent speech sound errors and distortions (apraxia of speech)
  * At least 2 of 3 of the following other features must be present:

    1. Impaired comprehension of syntactically complex sentences
    2. Spared single-word comprehension
    3. Spared object knowledge
* Global CDR® plus National Alzheimer's Coordinating Center Frontotemporal Lobar Degeneration (NACC FTLD) score of 0.5 or 1 during Screening.
* CDR® plus NACC FTLD language domain score of 0.5, 1 or 2 during Screening.
* Normal or corrected eyesight and auditory abilities, sufficient to perform all aspects of the study scales and assessments.
* Fluent in English, per Investigator judgement.
* Must have reliable study partner that is able to attend all study visits with participant. Study partner must be able to read, write, and understand the English language.

Exclusion Criteria:

* Brain Magnetic Resonance Image (MRI) incompatible with a diagnosis of nfvPPA.
* History or evidence of a central nervous system (CNS) condition other than nfvPPA which may cause symptoms of aphasia or dementia, including but not limited to Alzheimer's disease (AD), Dementia with Lewy Bodies (DLB), inflammatory/demyelinating CNS conditions, Creutzfeldt Jakob disease, vascular dementia, post-stroke dementia, etc.
* Features or Parkinsonism, corticobasal syndrome or progressive supranuclear palsy that are as or more prominent than the language features of nfvPPA, and/or motor features which are sufficiently severe that they could significantly impact performance on any of the clinical or neuropsychological measures.
* Plasma pTau217 result with a high likelihood of the presence of amyloid pathology at Screening or documented evidence of positive biomarkers associated with Alzheimer's disease pathology (e.g., abnormal plasma Aβ42/40 ratio, abnormal CSF phospo-tau/amyloid ratio, or presence of amyloid tracer update on brain amyloid positron emission tomography [PET] imaging).
* Known progranulin (GRN) mutations.
* Ongoing major and active psychiatric disorder and/or other concurrent medical condition that, in the opinion of the Investigator, might compromise safety and/or compliance with study requirements.
* Metabolic or toxic encephalopathy or dementia due to a general medical condition.
* History of previous neurosurgery to the brain within the past five years.
* Suicidality, defined as active suicidal thoughts within 6 months before Screening or at Baseline, defined as answering yes to items 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS), or history of suicide attempt in previous 2 years, or, in the Investigator's opinion, at serious risk of suicide.
* Clinically relevant intellectual impairment that may interfere with the ability to complete the study scales and assessments, at the discretion of the Investigator.
* Diagnosis of alcohol or drug abuse within the previous 2 years.
* Poorly controlled clinically significant medical illness, such as hypertension; myocardial infarction within 6 months; uncompensated congestive heart failure or other significant cardiovascular, pulmonary, renal, liver, infectious disease, immune disorder, or metabolic/endocrine disorders or other disease that would interfere with assessment of drug safety.
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2 × the upper limit of normal (ULN), total bilirubin >1.5 × ULN, and/or International Normalized Ratio (INR) >1.5.

  * If participant has a documented history of Gilbert's syndrome, criterion of total bilirubin >1.5 x ULN is not applicable.
  * If participant is taking anticoagulants (e.g., warfarin), and has no known liver issues, INR >3.
* Known human immunodeficiency virus, hepatitis B, or active hepatitis C virus infection.
* Participated in a study of an investigational drug or transcranial direct current stimulation less than 6 weeks or 5 half-lives of an investigational drug, whichever is longer, before enrollment in this study.
* Male with female partner(s) of childbearing potential, unwilling or unable to adhere to contraception requirements specified in the protocol.
* Female of childbearing potential (see Section 5.10), with a positive pregnancy test result during Screening and are unwilling or unable to adhere to contraception requirements specified in the protocol.
* Weight less than 50 kg at Screening.

The following additional exclusion criteria applies for participants undergoing (18F-Fluorodeoxyglucose Positron Emission Tomography-Computed Tomography) 18F-FDG PET-CT (18F-FDG PET-CT scans are optional):

* Blood glucose levels >200 mg/dL.
* Contraindications to having a PET scan.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events and Serious Adverse Events. | Baseline to Week 36
  The number and proportion of participants experiencing adverse events (AEs) and serious adverse events (SAEs) during the study period, categorized by severity and relationship to the study intervention.

OTHER OUTCOMES:
Change from Baseline to Week 36 in Digitized Speech Metrics | Baseline to Week 36
  Participant will complete a series of tasks in which voice recordings will be captures. The voice recording will be analyzed for linguistic and acoustic metrics.
Change from Baseline to Week 36 in Letter Fluency Test (LFT) | Baseline to Week 36
  The LFT is scored by counting the number of valid words a participant generates within a set time. Scores can range from 0 to 50. Higher scores indicate better verbal fluency and cognitive processing, while lower scores reflect difficulty in language, memory, and executive functioning.
Change from Baseline to Week 36 in Category Fluency Test (CFT) | Baseline to Week 36
  The CFT is scored by counting the number of valid words a participant generates with in a specific category in a set time. Higher scores indicate better semantic memory and executive functioning, while lower scores reflect impairments in cognitive processing or language abilities.
Change from Baseline to Week 36 in Stroop Color and Word Test (SCWT) | Baseline to Week 36
  The SCWT is scored based on the time taken to complete each of the four conditions and are scaled utilizing a norming method based upon participant age. Scaled scores range from 1 to 19. Faster times, and higher scaled scores, indicate stronger executive function.
Change from Baseline to Week 36 in Progressive Aphasia Severity Scale (PASS) | Baseline to Week 36
  The PASS is a tool for rating the presence and severity of symptoms across speech, language and functional communication domains in participants with progressive aphasia. Individual domain scores range from 0 (normal) to 3 (severe impairment). Each individual domain is summed to provide a PASS Sum of Boxes Score. A higher PASS Sum of Boxes Score indicates greater severity of symptoms.
Change from Baseline to Week 36 in Northwestern Anagram Test (NAT) | Baseline to Week 36
  The NAT examines non-verbal production of subject extracted wh-questions (SWh) and object extracted wh-questions (OWh). Scores for the NAT range from 0-10 (5 points each SWh- and OWh-Questions). A higher total score indicates better non-verbal sentence production, while a lower score reflects worse non-verbal sentence production.
Change from Baseline to Week 36 in Western Aphasia Battery-Revised (WAB-R) | Baseline to Week 36
  The WAB-R is a test designed to assess a participant's language impairment. The WAB-R measures both linguistic and non-linguistic skills. The core measure of aphasia is the Aphasia Quotient (AQ) and is derived from the Spontaneous Speech, Auditory Verbal Comprehension, Repetition, Naming and Word Finding section scores. The AQ can range from 0 to 100 with higher scores indicating milder language impairment and the lower scores indicating greater language impairment.
Change from Baseline to Week 36 in Clinical Dementia Rating Plus National Alzheimer's Coordinating Center Frontotemporal Lobar Degeneration Sum of Boxes (CDR® plus NACC FTLD-SB) | Baseline to Week 36
  The CDR® plus NACC FTLD is aimed at evaluating those suffering from or at risk for any of the forms of frontotemporal lobar degeneration. The CDR® plus NACC FTLD-SB is scored by summing ratings across 10 domains. Each domain is rated on a scale from 0 (no impairment) to 3 (serve impairment). The total score ranges from 0 to 30, where higher scores indicate greater cognitive and functional impairment.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Mayo Clinic, Rochester, Minnesota
  - The Ohio State University, Columbus, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No